CLINICAL TRIAL: NCT04197297
Title: Imaging Trial of Biomarkers to Guide Individualized Therapy in Patients With Brain Metastasis Receiving Radiotherapy
Brief Title: Brain Imaging Biomarkers in Patients With Brain Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-5380
Record Dates: First submitted 2019-11-25; First posted 2019-12-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Brain Metastases, Adult
Keywords: Radiation Therapy; Radiotherapy; Biomarkers; Magnetic Resonance Imaging; Computed Tomography; Radiosurgery
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Participants will undergo CT and MRIs before and after radiation therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT and MRI Scans (Other): Each patient will undergo a 3T MRI scan as well as a dynamic contrast-enhanced CT scan within one week prior to the start of treatment. Patients will also undergo a research 3T MRI scan and research dynamic contrast-enhanced CT scan at the one week post radiotherapy mark. An MRI scan during their 3 month post-treatment follow up visits will take place as per routine standard of care.
  Interventions: Diagnostic Test: CT and MRI Scans

INTERVENTIONS:
Diagnostic Test: CT and MRI Scans — CT and MRI scans will occur before and after radiation therapy.

SUMMARY:
A biomarker is a measurable indicator of the severity or presence of some disease state. In this study, brain metastases patients who will be receiving radiation treatment, will undergo CT (Computed Tomography) and MRI (Magnetic Resonance Imaging) scans prior to and after radiation treatment to measure these biomarkers. This is a single-center phase II study to validate the predictive abilities of biomarkers, in terms of determining how patients will respond to radiation treatment.

DETAILED DESCRIPTION:
Advances in medical imaging can provide useful information to guide and look at the response to treatment. Previous studies suggest early changes in the tumor after radiation treatment may be detectable using special MRI (Magnetic Resonance Imaging), and CT (Computed Tomography) scans. A biomarker is a measureable indicator of the severity or presence of some disease state. Previous studies suggest that the change in several imaging biomarkers can predict who will respond to radiation treatment. In this study, patients will undergo CT and MRI scans prior to and after radiation treatment to measure these biomarkers. The purpose of this study is to validate the predictive abilities of biomarkers in terms of determining how patients will respond to radiation treatment. This is a single-center phase II study, which will be conducted at the Princess Margaret Cancer Center. The study will be enrolling up to a total of 90 patients who will be receiving radiation treatment for brain metastases. Patients will be asked to participate within this study for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven primary malignancy (original biopsy is adequate as long as the brain imaging is consistent with brain metastases)
* At least one index lesion with diameter > 1cm and without imaging evidence of hemorrhage
* Patients age > 18 years of age
* Patients planned for RT to brain metastases
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Previous Whole Brain Radiotherapy
* Previous radiosurgery to the index lesion
* Individuals unable to undergo contrasted MRI for whatever reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Response Assessment in Neuro-Oncology (RANO) to validate biomarkers | Up to 2 years.
  Using RANO to validate imaging predictive biomarkers of response to radiotherapy
Response Evaluation Criteria in Solid Tumors (RECIST) criteria to validate biomarkers | Up to 2 years.
  Using RECIST criteria to validate imaging predictive biomarkers of response to radiotherapy
Progression Free Survival (PFS) to validate biomarkers | Up to 2 years.
  Using PFS to validate imaging predictive biomarkers of response to radiotherapy

SECONDARY OUTCOMES:
Objective (Radiological) Progression | Up to 2 years.
  Defined as increase in volume of contrast uptake on MRI of > 25% as measured by two perpendicular tumor diameters compared to the smallest measurement ever for the same lesion by the same technique.
Objective (Radiological) Response | Up to 2 years.
  Defined as stable or reduced volume of contrast uptake on MRI (i.e., all non-progression).
Time to Intracranial Local Progression | Up to 2 years.
  Defined as the time interval between the date of first treatment and the date of objective radiological progression of any one of the treated lesions.
Time to Intracranial Distant Progression | Up to 2 years.
  Defined as the time interval between the date of first treatment and the date of new brain metastases, with or without progression of the treated lesions.
Brain Progression Free Survival | Up to 2 years.
  Defined as the time interval between the date of first treatment and the date of disease progression in the brain or death due to disease in the brain, whichever comes first.
Unexpected and/or Serious Toxicities (AEs) | Up to 2 years.
  AEs that are deemed by the PI to be possibly, probably or definitely attributable to the research MRI and/or CT will be reported according to CTCAE version 4.3.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Coolens, Ph. D, Principal Investigator — Princess Margaret Cancer Center - UHN
Locations (1):
- University Health Network, Toronto, Ontario, Canada